CLINICAL TRIAL: NCT05981937
Title: Indocyanine Green ICG in Segmentary Resection in Colo-rectal Surgery is Usefull to Decrease Leak Threshold: A Paralel Retrospetive Cohort Study
Brief Title: ICG Anastomosis Control in Colon Surgery
Status: Completed | Type: Observational
Sponsor: Azienda Unita Sanitaria Locale di Piacenza (Other)
Responsible Party: Principal Investigator, Elena Orlandi, Principal Investigator, Medical Doctor, Azienda Unita Sanitaria Locale di Piacenza
Other Study IDs: GREEN COLONIC SAFE ANASTOMOSIS
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Colon Surgery; Anastomotic Leak
Keywords: ICG; Colon Surgery; Anastomotic Leak
MeSH Terms: conditions — Anastomotic Leak | interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Indocyanine Green: Indocyanine green infusion in left-side colorectal surgery (elective segmentary colic resection)
  Interventions: Drug: ICG solution
- non-Indocyanine Green: No infusion of Indocyanine green in left-side colorectal surgery (elective segmentary colic resection )

INTERVENTIONS:
Drug: ICG solution — ICG-ATT is available at our institute since 2019 using a near-infrared (NIR) light source and special scope and camera equipped with xenon light (CARL STORZ GmbH & Co. KG, Tuttlingen, Germany); ICG was supplied as a sterile water-soluble lyophilized powder (Diagnostic Green® GmbH). ICG-ATT is routinely used whenever available in daily practice with the following protocol: after the specimen resection the two colonic stumps or colonic and rectal stumps are checked with 5 cc of ICG 25 mg diluted in 10 cc of water sterile solution before fashioned anastomosis. Two laparoscopes with ICG-optic system are nowadays available department and ICG anastomosis control is always performed if ICG device are available (no performed in case of not available ICG instrument for sterilization in case of two consecutive surgery in the same day, concomitant ICG surgery or ICG malfunction).
  Other Names: Indocyanine Green
  Groups: Indocyanine Green

SUMMARY:
This is a parallel monocentric, retrospective cohort study in Guglielmo da Saliceto Hospital, Piacenza, Italy. Aim of this study is to investigate the protective role of Indocyanine green (ICG) for Anastomotic leak (AL) in patients underwent elective segmentary colic resection (transverse colic resection, left colectomy including sigmoidectomy, splenic colic flexure resection). Secondary aims are to detect and to investigate the impact of various risk factors on AL and morbidity and surgical performance within 30 days to surgery.

DETAILED DESCRIPTION:
This is a parallel monocentric, retrospective cohort study observing consecutive series of patients underwent colo-rectal surgery at our institution between 1 January 2017 and 31 July 2023.

The primary endpoint of the study is Anastomotic Leak (AL) at 30 days while secondary endpoints are post-operative morbidity Clavien-Dindo score ≥III within 30 days from surgery including readmission and redo-surgery, harvested nodes for patients with neoplastic disease, Surgical Site Infection, rate of laparoscopic surgical procedure and rate of protection stoma.

Sex, Body Mass Index, smoking, diabetes mellitus, cardiovascular disease, tumor stage according to AJJC 8th edition will be considered confounding factor for onset of AL.

Patients electronic database will be collected from extraction of medical record in operating log and every digital medical record will be scanned including peri-operative outcomes and 30 days post-operative follow-up from post-operative visit, eventually readmission in emergency department or any other specialistic wards of our local health institution according to following inclusion criteria: elective setting of surgery, segmentary left colon surgery: splenic colic resection, transverse colic resection and left colectomy defined as left hemicolectomy with low mesenteric artery-ligation and sigmoidectomy even for benign or malign pathology, at least 30 days of post-operative follow-up available from medical documentation, primary colo-colic or colo-rectal anastomosis with or without preventing ostomy and adult age.

Exclusion criteria are terminal colonic stoma without anastomosis creation after demolitive step, extended transverse right hemicolectomy, left hemicolectomy with high vascular ligation, associated bowel or another splanchnic resection (i.e. neoplastic infiltration), previous colic surgery, synchronous neoplasm, not reporting in operating form details about vascular ligation, lack in reporting in medical records of primary outcomes, stage IV cancer, ASA IV, less than 18 years old and emergency setting.

The reconstruction time is performed with different anastomosis (colo-colic or colo-rectal), technique (stapler or hand sewn) and connection (side to side, side to end, end to side or end to end).

ICG-ATT is available at our institute since 2019 using a near-infrared (NIR) light source and special scope and camera equipped with xenon light (CARL STORZ GmbH & Co. KG, Tuttlingen, Germany); ICG was supplied as a sterile water-soluble lyophilized powder (Diagnostic Green® GmbH). ICG-ATT is routinely used whenever available in daily practice with the following protocol: after the specimen resection the two colonic stumps or colonic and rectal stumps are checked with 5 cc of ICG 25 mg diluted in 10 cc of water sterile solution before fashioned anastomosis. Two laparoscopes with ICG-optic system are nowadays available department and ICG anastomosis control is always performed if ICG device are available (no performed in case of not available ICG instrument for sterilization in case of two consecutive surgery in the same day, concomitant ICG surgery or ICG malfunction).

Statistical analysis and sample size:

Quantitative variables will be described by mean± standard deviation or median and IQR, and qualitative variables will be described by absolute and percentage frequencies. Normality will be checked for all continuous variables. Comparisons of covariates will be conducted using Pearson's X2 test or Fisher's exact test for categorical variables and a t-test or Mann Whitney test for continuous variables. Univariable analysis will be conducted using logistic regression to examine the association of each predictor variable with the anastomotic leakage event. Next, variables with p<0.1 will be considered for inclusion in a multivariable regression model. For each risk factor, odds ratio with associated confidence intervals will have been presented. All analyses will be performed using RStudio version 3.6.0 statistical software with two-side significance tests and a 5% significance level.

ELIGIBILITY:
Inclusion criteria:

* elective setting of surgery
* segmentary left colon surgery including transverse resection, splenic flexure resection and left colectomy even for benign or malign pathology
* 30 days of post-operative follow-up at least available from medical documentation
* primary colo-colic or colo-rectal anastomosis with or without preventing ostomy
* more than 18 years old, less than 90 years old

Exclusion criteria:

* terminal colonic stoma without anastomosis creation after demolitive step
* extended transverse right hemicolectomy
* left hemicolectomy with high vascular ligation
* associated bowel or another splanchnic resection (i.e. neoplastic infiltration)
* previous colic surgery
* synchronous neoplasm
* not reporting in operating form details about vascular ligation
* lack in reporting in medical records of primary outcomes
* stage IV cancer
* ASA IV
* less than 18 years old, more then 90 years old
* emergency setting

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive series of patients underwent colo-rectal surgery at our institution between 1 January 2017 and 31 July 2023
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Anastomotic leak at 30 days | 30 days
  Anastomotic leak (a defect of intestinal wall at anastomotic site leading to a communication between the intra- and extraluminal compartments)at 30 days: abdominal CT scan IV and a Clavien Dindo Score ≥III

SECONDARY OUTCOMES:
Post-operative morbidity | 30 days
  Clavien-Dindo score ≥III within 30 days from surgery including readmission and redo-surgery, harvested nodes for patients with neoplastic disease, Surgical Site Infection, rate of laparoscopic surgical procedure and rate of protection stoma.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Romboli, MD, Principal Investigator
Locations (1):
- Guglielmo da Saliceto Hospital, Piacenza, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Romboli A, Orlandi E, Citterio C, Banchini F, Ribolla M, Palmieri G, Giuffrida M, Luzietti E, Capelli P. Indocyanine green in left side colorectal surgery segmental resection to decrease anastomotic leak: A parallel retrospective cohort study of 115 patients. Heliyon. 2024 Oct 24;10(23):e39730. doi: 10.1016/j.heliyon.2024.e39730. eCollection 2024 Dec 15. PMID 39687188